CLINICAL TRIAL: NCT05863546
Title: Effect of Different Doses of Therapeutic Ultrasound in the Treatment of Carpal Tunnel Syndrome
Brief Title: Effect of Different Doses of US in the Treatment of CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Gamal Mohamed, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003996
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Sham Comparator): (control group) It consisted of 15 subjects who received a program of 'sham' US application, so that the US device was working but not delivering any output plus traditional PT treatment for carpal tunnel syndrome which included hot packs, tendon glide and nerve glide exercises, US treatment sessions were performed for 6 min per session, once a day, three days a week, for a total of 4 weeks.
  Interventions: Other: Traditional treatment; Device: Therapeutic ultrasound
- Low-dose group (Experimental): (low-dose group) It consisted of 15 subjects who received a program of US treatments that was administered to the carpal tunnel area with pulsed mode at a frequency of 1 MHz with an intensity of 0.25 W/cm2 and a duty cycle of 1:4 plus traditional treatment.
  Interventions: Other: Traditional treatment; Device: Therapeutic ultrasound
- Mid-dose group (Experimental): (Mid-dose group) It consisted of 15 subjects who received a program of US treatments that was administered to the carpal tunnel area with pulsed mode at a frequency of 1 MHz with an intensity of 0.5 W/cm2 and a duty cycle of 1:4 plus traditional treatment.
  Interventions: Other: Traditional treatment; Device: Therapeutic ultrasound
- High-dose group (Experimental): (high-dose group) It consisted of 15 subjects who received a program of the same US equipment that was set at pulsed mode at a frequency of 1 MHz, intensity of 1.0W/ cm2 and a duty cycle of 1:4 plus traditional treatment.
  Interventions: Other: Traditional treatment; Device: Therapeutic ultrasound

INTERVENTIONS:
Other: Traditional treatment — The patients received traditional physical therapy treatment for carpal tunnel syndrome, in the form of hot packs, tendon and nerve glide exercises, and wrist splint for 4 weeks.
Device: Therapeutic ultrasound — US treatment sessions were performed for 6 min per session, once a day, three days a week, for a total of 4 weeks.

SUMMARY:
The purpose of this study was to investigate the effective dose of therapeutic ultrasound in the treatment of carpal tunnel syndrome on pain level, functional ability, motor and sensory nerve conduction parameters and pinch strength.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is among the most common peripheral neuropathies causing the median nerve compression as it crosses the carpal tunnel, with an estimated prevalence of about 4 - 5% of the general population. Patients suffering from this syndrome mainly complain about paresthesia (pain, numbness, and tingling) in the innervation area of the median nerve in the hand which could be accompanied by weakness and atrophy of thenar muscles.

Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy of the upper limb and a significant contributor to hand functional impairment and disability that could be treated through numerous approaches. Effective treatment options include conservative and surgical interventions.

Carpal Tunnel Syndrome (CTS) remains a puzzling and disabling condition present in 3.8% of the general population. CTS is the most well-known and frequent form of median nerve entrapment, and accounts for 90% of all entrapment neuropathies.

Physiotherapy modalities are used to help patients with CTS in many cases. They can both help to improve CTS symptoms as well as resolve the cause of the syndrome. Physiotherapy intervention may include special exercises, mobilizations, ergonomic interventions and advice for as well as electrotherapy modalities, aiming for the treatment and improvement of symptoms.

Ultrasound waves have anti-inflammatory properties, stimulating nerve regeneration and improving nerve conductivity.

The most common uses for US are to decrease soft tissue inflammation, increase tissue extensibility, enhance scar tissue remodeling, increase soft tissue healing, decrease pain, and decrease soft tissue swelling .

The issue of selecting the nature of the ultrasonic wave has not been finally resolved. A continuous wave is more often used to reduce pain and increase the elasticity of the tissue, while a pulsed wave mode is applied to reduce swelling and to eliminate inflammation. The rate of absorption, and thus the thermal effect, is based on the tissue type encountered, the frequency of the ultrasound beam, and the intensity (W/cm2) of the ultrasonic output.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age range was 25-55 years .
2. Mild to moderate CTS, that is confirmed by neurologist or orthopedist based on results of physical examination and electrophysiological criteria; i. Mild CTS is characterized by sensory fibers involvement (sensory peak latency > 3.6 milliseconds) with no motor fiber involvement (motor distal latency < 4.1 milliseconds), provided that sensory nerve action potential (SNAP) is not absent.

   ii. Moderate CTS is characterized by involvement of both sensory and motor fibers, provided that neither of these two waves is absent .
3. Pain intensity more than 5 in visual analogue scale (VAS).

Exclusion Criteria:

1. History of any trauma on the hands, neck, and shoulders within 3 months of the study onset
2. Cervical radiculopathy, peripheral polyneuropathy, or other neurological conditions.
3. Patients suffering from severe CTS according to electrophysiological criteria

   -

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
symptoms severity and functional status | Four weeks
  Symptoms severity and functional status were measured by Boston carpal tunnel syndrome questionnaire. The patients rated their ability to perform the activity on a scale that ranged from 1 (no difficulty with the activity) to 5 (cannot perform the activity at all).
median nerve motor distal latency | Four weeks
  Electrodiagnostic tests were used to measure median nerve motor distal latency in milliseconds.
median nerve motor amplitude | Four weeks
  Electrodiagnostic tests were used to measure motor amplitude in millivolt.
median nerve sensory distal latency | Four weeks
  Electrodiagnostic tests were used to measure median nerve sensory distal latency in milliseconds.
median nerve sensory amplitude | Four weeks
  Electrodiagnostic tests were used to measure sensory amplitude in millivolt
Pain intensity | Four weeks
  Pain intensity was measured by visual analogue scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Pinch strength | Four weeks
  Pinch dynamometer was used to measure pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Ragia Mohamed Kamel, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Ismailia Medical Complex, Ismailia, Egypt